CLINICAL TRIAL: NCT02284711
Title: Impact of Salpingectomy on Ovarian Reserve, With Comparison Between Two Coagulation Techniques
Brief Title: Impact of Salpingectomy on Ovarian Reserve
Acronym: SALPOVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69HCL14_0166; 2014-A01218-39 (Other: ID-RCB)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Laparoscopic Salpingectomy
Keywords: salpingectomy, ovarian reserve, coagulation technique
MeSH Terms: interventions — Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bipolar (Active Comparator): Coagulation during salpingectomy using conventional bipolar electric energy
  Interventions: Device: Bipolar electric energy
- Ultrasound (Active Comparator): Coagulation during salpingectomy using UltraCision HARMONIC ACE® ultrasound energy
  Interventions: Device: ultrasound energy

INTERVENTIONS:
Device: Bipolar electric energy — Coagulation during salpingectomy using conventional bipolar electric energy
  Arms: Bipolar
Device: ultrasound energy — Coagulation during salpingectomy using UltraCision HARMONIC ACE® ultrasound energy
  Arms: Ultrasound

SUMMARY:
Epithelial cancer of the ovaries is the most severe form of gynecologic cancer; a significant proportion of ovarian cancers originate from the Fallopian tube. Guidelines therefore now recommend systematically associating prophylactic salpingectomy to benign hysterectomy. The principal objective of the present study is to assess the impact of salpingectomy on ovarian reserve by anti-Müllerian hormone (AMH) assay and calculating the Doppler index of vascular resistance in the ovarian vessels. The secondary objective is to compare ovarian reserve results between two coagulation techniques used in salpingectomy: bipolar electric energy versus ultrasound.

The study design is single-center, prospective, before-and-after, with open randomization between two groups defined by coagulation technique.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged 18
* Scheduled surgery: bilateral laparoscopic salpingectomy associated to hysterectomy for benign indication

Exclusion Criteria:

* Interview revealing disorder entailing unacceptable risk of postoperative complications: coagulation disorder, immune system disorder, evolutive disease, etc.
* Pregnancy, ongoing or planned during the study period
* History of bilateral salpingectomy
* Salpingectomy associated with pelvic cancer
* Oral hormonal contraception during the study period
* Menopause
* Inability to understand information provided
* Not covered by a national health insurance scheme, prisoner or under administrative supervision.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
AMH level | 3 months post-surgery

SECONDARY OUTCOMES:
AMH level | 1 month post-surgery
index of vascular resistance in the ovarian vessels | 1 and 3 months post-surgery
menopausal quality of life score | 1 and 3 months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - HFME, Lyon, France

REFERENCES:
- [Background] Lamblin G, Thiberville G, Bansac Lamblin A, Moret S, Du-Mesnildot P, Rannou C, Ploton I, Chabert P, Chene G. [What haemostatic technique should we use for opportunistic salpingectomy during benign laparoscopic hysterectomy?]. Gynecol Obstet Fertil Senol. 2017 Sep;45(9):453-459. doi: 10.1016/j.gofs.2017.06.017. Epub 2017 Jul 27. French. PMID 28757104